CLINICAL TRIAL: NCT03934658
Title: A Remote Randomized Double-Blind Sham-Controlled Clinical Trial of NightWare in Adults With Post-Traumatic Stress Disorder and Co-Morbid Nightmare Disorder
Brief Title: Remote Study of NightWare for PTSD With Nightmares
Acronym: NWVRCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NightWare (Industry)
Collaborators: RationalPsych (Unknown); Center for International Emergency Medical Services (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NW101004
Record Dates: First submitted 2019-04-29; First posted 2019-05-02 (Actual); Last update posted 2022-01-28 (Actual); Status verified 2022-01

CONDITIONS: PostTraumatic Stress Disorder; Sleep Disorder; Stress Disorder; Sleep Initiation and Maintenance Disorders; Combat Disorders; Nightmares Associated With Chronic Post-Traumatic Stress Disorder; Nightmare; Nightmares, REM-Sleep Type
Keywords: PTSD; Nightmare Disorder; Post-traumatic stress disorder; Veteran; Digital therapeutic; Digital medicine; Nightmares
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Sleep Wake Disorders; Stress Disorders, Traumatic; Sleep Initiation and Maintenance Disorders; Combat Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Active Treatment Arm (Experimental): Intervention with the NightWare Therapeutic System every night.
  Interventions: Device: NightWare Therapeutic System
- Sham Arm (Sham Comparator): NightWare Therapeutic System every night with interventions not-enabled.
  Interventions: Device: NightWare Therapeutic System in Sham Mode

INTERVENTIONS:
Device: NightWare Therapeutic System — A wearable digital therapeutic system that will measure physiologic data when worn during sleep to deliver a mild vibration via the watch to elicit arousal thereby disrupting nightmares. This detection and stimulation sequence will be performed according to NightWare's proprietary algorithm.
  Arms: Active Treatment Arm
Device: NightWare Therapeutic System in Sham Mode — A wearable digital therapeutic system that will measure physiologic data when worn during sleep that does not deliver interventions.
  Arms: Sham Arm

SUMMARY:
This study will provide measures of safety and efficacy of the NightWare digital therapeutic system (iPhone + Apple watch + proprietary application) for the treatment of nightmare disorder associated with post-traumatic stress disorder (PTSD)-related sleep disturbance and the impact of improved sleep with the NightWare digital therapeutic system. The investigators hypothesize that the NightWare digital therapeutic system will significantly improve sleep quality in participants with PTSD-Related nightmares and poor sleep quality.

DETAILED DESCRIPTION:
Nightmares are a common problem affecting 2-8% of the general population and a higher proportion of clinical populations. The negative consequences of untreated nightmares are significant and include impaired quality of life, sleep deprivation (often resulting in an increased intensity of nightmares), insomnia, daytime sleepiness, and fatigue. Untreated nightmares can also exacerbate the symptoms of underlying psychological dysfunction in people with depression and anxiety, leading to poor occupational and or social functioning. Nightmares can be idiopathic or associated with the use (or withdrawal) of certain medications or substances or associated with disorders including PTSD.

NightWare (Minneapolis, MN) has developed a novel approach to the treatment of nightmares. Through the use of a smartwatch-based application that senses physiologic parameters, the participant is aroused from sleep (without awakening the participant) so that the nightmare is interrupted prior to reaching a threshold of severity in which the participant would awaken in distress. Seconds later the participant returns to sleep without having experienced a nightmare. This approach avoids risk from pharmacological treatment, avoids exacerbation of symptoms from image rehearsal therapy and allows for a simple method with easily achieved adherence compared to existing treatments.

The NightWare digital therapeutic system consists of a proprietary software application installed on a smartwatch. The application has been effective in focus groups when used on both Apple smartwatches and Motorola smartwatches. For the purposes of this study, the investigators will be using only the Apple (Cupertino, CA) 3rd generation smartwatch and the Apple iPhone. The NightWare application uses physiological markers obtained via the smartwatch to determine by proprietary algorithm whether a participant is in the early stages of a nightmare, but has not yet awoken in distress. As directed by the algorithm, the smartwatch then applies varying degrees of vibratory stimulation to the wrist over variable lengths of time with the intention of arousing the participant from sleep without eliciting an awakening.

ELIGIBILITY:
Inclusion Criteria

* Self report of diagnosis with PTSD
* Self-report of PTSD-related repetitive nightmares contributing to disrupted sleep.
* Equal to or older than 18 years of age.
* Proficient in both reading and writing in the English language.
* Pittsburgh Sleep Quality Index (PSQI) score equal to or greater than 10.
* ESS: On question #8 any score above "0" will prompt an additional question:
* Do you drive ("get behind the wheel") when you are drowsy? Answer must be "No" to be enrolled in the study for safety.
* Participant owns or has access to devices appropriate for participation in the study including compatible Apple Watch and Apple iPhone.
* Wireless Internet and two power outlets where they sleep.
* Willingness not to use any other application which collects heart rate data on the phone and watch that is used for NightWare.

Exclusion Criteria

* Circadian rhythm disruption on a regular basis (shift-work)
* Concurrent presence of prohibited medications
* Current use of varenicline
* Current use of beta-blockers (unless ophthalmic solutions)
* Current use of non-dihydropyridines
* Current use of Prazosin for the treatment of nightmares (can include subjects 2 weeks post-taper and discontinuation)
* Concurrent presence of prohibited diagnoses
* Known diagnosis of OSA
* Diagnosis of an active disorder of arousal from non-rapid eye movement sleep
* Diagnosis of rapid eye movement sleep behavior disorder
* Diagnosis of narcolepsy
* Diagnosis of dementia
* Uncontrolled atrial fibrillation
* Use of Alcohol or Drugs as specified:
* Alcohol Use Disorders Inventory Test (AUDIT) (score of 8 or higher)
* Drug Abuse Screening Test-10 (DAST-10) (score greater than 2)
* Suspicion of nightmares being secondary to substance abuse or withdrawal
* Previous or foreseeable legal proceedings involving nightmares or trauma
* Nocturia that causes awakening from sleep
* Known sleep walking
* Acting out of dreams PRIOR to PTSD trauma
* Self reported pregnancy or intent to become pregnant during the course of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2019-05-21 (Actual); Primary Completion 2021-12-15 (Actual); Study Completion 2021-12-15 (Actual)

PRIMARY OUTCOMES:
Change in global score on the Pittsburgh Sleep Quality Index (PSQI) from Day 0 to each subsequent 28 day evaluation period | 0-730 days
  The Pittsburgh Sleep Quality Index (PSQI) is a self-rated questionnaire which assesses sleep quality and disturbances over a 1-month time interval. Nineteen individual items generate seven "component" scores: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction. The sum of scores for these seven components yields one global score. In scoring the PSQI, seven component scores are derived, each scored 0 (no difficulty) to 3 (severe difficulty). The component scores are summed to produce a global score (range 0 to 21). Higher scores indicate worse sleep quality. This outcome is the difference between the global score on the Pittsburgh Sleep Quality Index (PSQI) score at baseline (Day 0) and average global PSQI score across the post-treatment initiation assessments (Days 14, 28 and every 28 days after that).

CONTACTS AND LOCATIONS:
Overall Officials: Daniel R Karlin, MD MA, Principal Investigator — RationalPsych
Locations (1):
- RationalPsych, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: Yes